CLINICAL TRIAL: NCT03924440
Title: Characterization and Use of Urine Pregnanediol Rapid Test and Its Use for Confirming Ovulation - Proov (Ovulation Double Check) Test
Brief Title: Ovulation Double Check (Proov) Verification and Usability Testing
Status: Completed | Type: Observational
Sponsor: MFB Fertility (Industry)
Responsible Party: Sponsor
Other Study IDs: 09/19/2016
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ovulation Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PDG Test strip Users: Participants were asked to predict ovulation by monitoring changes in cervical mucus and/or tracking luteinizing hormone (LH) via home test kits. Participants were asked to self-report their peak fertility day, which was defined as the first LH surge day and/or day of peak cervical mucus (stretchy and eggwhite in consistence).
  Participants collected first morning urine as various times during their cycle, including, prior to, during, and after peak fertility signs were observed. Participants were provided PDG rapid response test strips and self-administered their tests and recorded their results. Test results were reported back researchers via a log sheet. Log sheets recorded testing date, day of cycle, date of peak fertility (if known), personal assessment of results (positive result vs negative result) and a place to tape the completed test strip.
  Interventions: Diagnostic Test: Proov (Ovulation Double Check) Test

INTERVENTIONS:
Diagnostic Test: Proov (Ovulation Double Check) Test — Rapid response urine progesterone test strips, Proov (formerly named Ovulation Double Check

SUMMARY:
The Ovulation Double Check test is a Class I, 510K exempt medical device. It is manufactured and packaged in an FDA-registered and cGMP compliant facility. This device measures the level of Pregnanediol (PdG), the major urine metabolite of progesterone, in the urine of women. PdG has been shown to increase significantly after ovulation has occurred. This test will be used in a home setting as a point-of-care device, providing couples additional information about menstrual cycling and possible fertile periods. The investigators have successfully developed prototype devices that can accurately measure PdG in urine. Now the investigators need to supply these prototype devices to end users to verify the assay is working correctly and determine if the device was designed properly in order for home users to 1) use the test properly, 2) read the test results properly, and 3) interpret the results correctly.

DETAILED DESCRIPTION:
Lack of or insufficient ovulatory events is the primary cause of infertility worldwide and with 12% of couples within the US being diagnosed with infertility each year (according to the CDC), thus being able to confirm ovulation is an essential component of infertility evaluations in women. The gold standards for confirming ovulation include transvaginal ultrasounds and serum progesterone blood draws. Both of these techniques are too invasive, too expensive, and/or inaccessible to most women. Therefore a non-invasive, inexpensive, home-based testing system to confirm ovulation is desired. Several recent studies have identified urinary pregnanediol levels as an accurate way to confirm ovulation. However, until now, urine pregnanediol levels were always measured via a lab setting. Here the investigators describe the development of a urine pregnanediol (PDG) rapid test and its use at confirming ovulation in a home environment. Study Protocol One hundred and ninety six women were recruited to take part in a prospective, blinded cohort home environment study. The study protocol was approved by the Ethics Committee at Solutions IRB. Detailed information about the study was provided to each volunteer, and informed consent was obtained prior the study commencement. Inclusion criteria were non-pregnant women residing within the United States, aged 18- 45, and not currently on hormonal birth control. Importantly, women were not excluding due to average cycle length, weight (BMI), breastfeeding status, poly-cyctic ovarian syndrome (PCOS) or any other cause of infertility or lifestyle factor. Participants were asked to predict ovulation by monitoring changes in cervical mucus and/or tracking luteinizing hormone (LH) via home test kits. Participants were asked to self-report their peak fertility day, which was defined as the first LH surge day and/or day of peak cervical mucus (stretchy and eggwhite in consistence).

Participants collected first morning urine as various times during their cycle, including, prior to, during, and after peak fertility signs were observed. Participants were provided PDG rapid response test strips and self-administered the tests and recorded the results. Test results were reported back the investigators via a log sheet. Log sheets recorded testing date, day of cycle, date of peak fertility (if known), personal assessment of results (positive result vs negative result) and a place to tape the completed test strip.

ELIGIBILITY:
Inclusion Criteria:

1. Female (mandatory)
2. Not currently pregnant or nursing (pregnancy affects PdG levels)
3. Aged 18-34 (advanced age can hinder PdG levels)
4. Cycle length of 26-39 days (long or short cycles have inconsistent PdG levels)
5. Currently use other fertility monitoring tools (this allows us to compare Proov - Ovulation Double Check test results with other fertility tracking methods)

Exclusion Criteria:

1. Male
2. Pregnant
3. Nursing

Ages: 18 Years to 34 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Women only due to ovulation tracking diagnostic studied
Study Population: Inclusion criteria were non-pregnant women residing within the United States, aged 18-34, and not currently on hormonal birth control. Importantly, women were not excluding due to average cycle length, weight (BMI), breastfeeding status, poly-cyctic ovarian syndrome (PCOS) or any other cause of infertility or lifestyle factor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number if participants with positive PDG test results | A single menstrual cycle, up to 45 days.
  PDG test results are recorded to determine when PDG test results were positive

CONTACTS AND LOCATIONS:
Overall Officials: Amy Beckley, PhD, Principal Investigator — MFB Fertility

IPD SHARING:
Plan to Share IPD: No